CLINICAL TRIAL: NCT00677898
Title: A Patient-Centered Approach to Improve Screening for Side Effects of SGAs
Brief Title: A Patient-Centered Approach to Improve Screening for Side Effects of Second Generation Antipsychotics (SGAs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-256
Record Dates: First submitted 2008-05-09; First posted 2008-05-15 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-08

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Patient-Centered Care; Adverse effects; Antipsychotics
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient-centered computerized tool (Experimental): A brief computer program that provides personalized health information to patients prescribed second-generation antipsychotic medications on adherence to guidelines for screening of metabolic side effects
  Interventions: Behavioral: Patient-centered computerized tool
- Written educational materials (Active Comparator): Printed information on the metabolic side effects of second-generation antipsychotic medications and general recommendations for screening
  Interventions: Behavioral: Written educational materials

INTERVENTIONS:
Behavioral: Patient-centered computerized tool — A brief computer program that provides personalized health information to patients prescribed second-generation antipsychotic medications on adherence to guidelines for screening of metabolic side effects
  Arms: Patient-centered computerized tool
Behavioral: Written educational materials — Printed information on the metabolic side effects of second-generation antipsychotic medications and general recommendations for screening
  Arms: Written educational materials

SUMMARY:
The purpose of this study is to determine if individuals with serious mental illnesses exposed to a patient-centered computerized tool versus printed educational materials have higher rates of screening for the metabolic side effects of second-generation antipsychotic medications and different patterns of communication with their prescribers about screening.

DETAILED DESCRIPTION:
Project Background/Rationale: Second-generation antipsychotic (SGA) medications are widely used to treat psychotic disorders but are associated with metabolic side effects such as weight gain, glucose dysregulation, and hyperlipidemia that may contribute to the high rates of cardiovascular disease observed in individuals with serious mental illness (SMI). Adherence to guidelines for regular screening for the metabolic side effects of SGAs is inadequate. Patient-centered care, characterized by an effective partnership between clinicians and patients that promotes active participation by patients in their own care, improves health outcomes and satisfaction in the general population. In order to increase rates of screening for the metabolic side effects of SGAs, we propose to design a patient-centered computerized tool that provides veterans with SMI with personalized health information on how well their care adheres to screening recommendations. The computerized tool will use principles shown to enhance usability in persons with cognitive impairments.

Project Objectives: The objectives of this study are to determine the effect of exposure to a patient-centered computerized tool compared to enhanced treatment as usual (e-TAU) on: (1) rates of screening for and identification of health problems associated with the metabolic side effects of SGAs; (2) patterns of patient-centered communication around screening for metabolic side effects and VA patients' self-efficacy in communicating with their psychiatrists about screening; (3) VA patients' preferences for obtaining health information and participating in decision-making about screening; and (4) VA patients' perceptions of their psychiatrists' participatory decision-making styles around screening.

Project Methods: A total of 240 veterans with psychotic disorders prescribed SGAs and in regular contact with their prescribing clinicians in outpatient mental health clinics in the VA Maryland Health Care System will be recruited for this randomized controlled trial. Half of participants will be randomly assigned to the intervention condition in which they will view a brief computer program that provides personalized health information on adherence to guidelines for screening of metabolic side effects that is designed to facilitate discussion with psychiatrists about appropriate screening. The other half of participants will receive enhanced treatment-as-usual (e-TAU) consisting of printed information on the metabolic side effects of SGAs and general recommendations for screening. Participants will be exposed to the intervention or e-TAU up to 3 times immediately prior to a visit with their prescriber over the one-year study period. Rates of screening for the metabolic side effects of SGAs will be obtained from patients' computerized medical records. A single prescriber visit for each participant will be audiotaped and coded with the Roter Interaction Analysis System (RIAS) to characterize patterns of patient-clinician communication around screening for metabolic side effects. Baseline and 12-month follow-up interview assessments with veterans will be used to acquire information on self-efficacy, their preferences for obtaining health information and participating in decisions regarding side effect screening, and important covariates such as severity of psychiatric illness.

ELIGIBILITY:
Inclusion Criteria:

* Agreement obtained from the treating clinician that the patient is clinically stable enough to participate in the study and can be contacted for recruitment
* Agreement obtained from treating clinician to have a single visit with the patient audio taped
* Patient age 18-70 years
* Diagnosis of a psychotic disorder (schizophrenia, affective psychosis, major depression with psychotic features)
* Currently prescribed any SGA medication (aripiprazole, clozapine, olanzapine, quetiapine, risperidone, ziprasidone) by a clinician in a VA Maryland Healthcare System (VAMHCS) mental health clinic
* Had at least two outpatient visits with the prescribing clinician in the past year - Decisional capacity to provide informed consent
* Ability to read at a 4th grade reading level

Exclusion Criteria:

* Diagnosis of dementia or other organic brain syndrome or traumatic brain injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Anne Kreyenbuhl, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

REFERENCES:
- [Result] Park SG, Derman M, Dixon LB, Brown CH, Klingaman EA, Fang LJ, Medoff DR, Kreyenbuhl J. Factors associated with shared decision-making preferences among veterans with serious mental illness. Psychiatr Serv. 2014 Dec 1;65(12):1409-13. doi: 10.1176/appi.ps.201400131. Epub 2014 Nov 17. PMID 25178383

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials
Started | 119 | 120
Completed | 99 | 102
Not Completed | 20 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials | Total
Number analyzed (Participants) | 119 | 120 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (8.0) | 53.5 (8.6) | 54.3 (8.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 116 | 227
  >=65 years | 8 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 107 | 106 | 213
Region of Enrollment [Number; unit: participants]
  United States | 119 | 120 | 239

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days in the Study Period That a Patient's Screening for Metabolic Side Effects of Second-generation Antipsychotic Medications Adheres to Guidelines: Body Mass Index
Description: Guidelines recommend that body mass index be evaluated every 3 months
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of days in the study period
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials
Number analyzed (Participants) | 119 | 120
percentage of days in the study period | 81.4 (22.5) | 76.1 (26.2)

2. Primary Outcome: Percentage of Days in the Study Period That a Patient's Screening for Metabolic Side Effects of Second-generation Antipsychotic Medications Adheres to Guidelines: Blood Pressure
Description: Guidelines recommend that blood pressure be evaluated every 3 months
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of days in the study period
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials
Number analyzed (Participants) | 119 | 120
percentage of days in the study period | 83.5 (21.8) | 78.5 (27.5)

3. Primary Outcome: Percentage of Days in the Study Period That a Patient's Screening for Metabolic Side Effects of Second-generation Antipsychotic Medications Adheres to Guidelines: Blood Glucose/HbA1c
Description: Guidelines recommend that blood glucose/HbA1c be evaluated every year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of days in the study period
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials
Number analyzed (Participants) | 119 | 120
percentage of days in the study period | 97.7 (10.7) | 96.2 (14.8)

4. Primary Outcome: Percentage of Days in the Study Period That a Patient's Screening for Metabolic Side Effects of Second-generation Antipsychotic Medications Adheres to Guidelines: LDL Cholesterol
Description: Guidelines recommend that LDL cholesterol be evaluated every 2 years
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of days in study period
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials
Number analyzed (Participants) | 119 | 120
percentage of days in study period | 93.7 (17.0) | 95.1 (14.3)

5. Primary Outcome: Percentage of Days in the Study Period That a Patient's Screening for Metabolic Side Effects of Second-generation Antipsychotic Medications Adheres to Guidelines: HDL Cholesterol
Description: Guidelines recommend that HDL cholesterol be evaluated every 2 years
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of days in study period
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials
Number analyzed (Participants) | 119 | 120
percentage of days in study period | 94.1 (16.6) | 95.2 (14.3)

6. Primary Outcome: Percentage of Days in the Study Period That a Patient's Screening for Metabolic Side Effects of Second-generation Antipsychotic Medications Adheres to Guidelines: Triglycerides
Description: Guidelines recommend that triglycerides be evaluated every 2 years
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of days in the study period
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials
Number analyzed (Participants) | 119 | 120
percentage of days in the study period | 94.1 (16.6) | 94.5 (15.1)

ADVERSE EVENTS:
Arm/Group | Patient-centered Computerized Tool | Written Educational Materials
Serious Adverse Events (participants affected / at risk) | 2/119 | 2/120
Other Adverse Events (participants affected / at risk) | 0/119 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient-centered Computerized Tool (N=119) | Written Educational Materials (N=120)
Death (General disorders) | 2 (2) | 2 (2) — All deaths that occurred during the study were reported to the local Institutional Review Board (IRB) and were determined to be unrelated to study participation.
Psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — All psychiatric hospitalizations that occurred during the study were reported to the local Institutional Review Board (IRB) and were determined to be unrelated to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes